CLINICAL TRIAL: NCT06390293
Title: The Effectiveness of Group-Delivered Revised Written Exposure Therapy for PTSD and Subclinical PTSD Among Chinese Adolescents: A Randomized Controlled Trial
Brief Title: The Effectiveness of Group-Delivered Revised Guided Written Exposure Therapy for PTSD and Subclinical PTSD Among Chinese Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, Research Fellow, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Guided WET-R on adolescents
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: PTSD
Keywords: PTSD; written exposure therapy; randomized controlled trial; adolescents
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group guided WET-R (Experimental)
  Interventions: Behavioral: Group-delivered guided written exposure therapy-revised version
- Waiting-List (WL) condition (Other)
  Interventions: Behavioral: Waiting-List (WL) condition

INTERVENTIONS:
Behavioral: Group-delivered guided written exposure therapy-revised version — Group-Delivered guided WET-R is a manualized exposure-based therapy program consisting of 5-8 sequential sessions. The interval between every 2 consecutive sessions is 0-2 days. There will be 5-8 group-delivered sessions in total (only one index trauma will be discussed), and 1-2 weeks to complete. The first and last sessions are scheduled to last for 1.5 hours each, while the other sessions will be 50 minutes in duration.
  Arms: Group guided WET-R
Behavioral: Waiting-List (WL) condition — Participants assigned to WL will be asked to not work with other therapists or seek additional treatment for trauma-related difficulties during the 2-week WL period. After the one-month follow-up of the WET-R group, they will receive the same treatment (Group-Delivered guided written exposure therapy-revised version).WL participants will also be given contact information to use in case of worsening symptoms or increasing distress.
  Arms: Waiting-List (WL) condition

SUMMARY:
The study aims to examine the effectiveness of the group-delivered revised written exposure therapy (WET-R) for post-traumatic stress disorder (PTSD) and subclinical PTSD among Chinese adolescents with a randomized controlled trial. The study will recruit 70 participants, with 35 randomized to the WET-R group and 35 randomized to the waiting list (WL) group. The WET-R intervention consists of 5-8 group sessions. The primary outcome CPSS-5-I (Child PTSD Symptom Scale-Interview Version for DSM-5) and PCL-5 ( PTSD Checklist-5) will be administered on baseline, post-treatment, 1-month follow-up, 3-month follow-up, and 6-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 10-18 years.
2. Meeting full or subthreshold PTSD (up to one symptom missing) diagnostic criteria according to the Child PTSD Symptom Scale-Interview Version for DSM-5 (CPSS-5-I).
3. If taking psychotropic medication, currently stabilized on psychotropic medication for at least four weeks.
4. Capable of writing and understanding written instructions.

Exclusion Criteria:

1. Presence of severe psychopathology necessitating immediate medical attention
2. Moderate to high suicide risk (e.g., intent or plan to attempt suicide in the near future
3. Evidence of a moderate or severe traumatic brain injury
4. Currently undergoing psychotherapy specifically for PTSD.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist-5 (PCL-5) | baseline,post treatment(2 weeks), 6 weeks, 14 weeks, 26 weeks
  PCL-5 was a 20-item self-report scale that assesses PTSD DSM-5 diagnosis and symptom severity in the past month. Items were rated on a 5-point Likert scale from 0 ("not at all") to 4("extremely").The Chinese version of PCL-5 has shown good psychometric properties in trauma-affected Chinese children.
Child PTSD Symptom Scale-Interview Version for DSM-5 (CPSS-5-I) | baseline,post treatment(2 weeks), 6 weeks, 14 weeks，26 weeks
  The PTSD Symptom Scale, CPSS-5-I is a 27-item semi-structured interview that assesses PTSD DSM-5 diagnosis and symptom severity in the past month based on interviewer ratings. The CPSS-5-I assesses history of Criterion A traumatic experiences to identify an index trauma.The 20 items assessing DSM-5 PTSD symptoms are presented. The interviewer rates each item from 0 (not at all) to 4 (6 or more times a week/almost always) based on the frequency and severity of the reported symptom experienced in the past month related to the index trauma. Finally, seven items assess impairment of endorsed symptoms on daily functioning pertinent to youth. The interviewer rates these items on a scale of 0 (not at all) to 4( 6 or more times a week/almost always).The total impairment score does not contribute to the overall severity score.CPSS-5-I has demonstrated excellent reliability and validity .

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided